CLINICAL TRIAL: NCT04514445
Title: Bicuspid aoRtic vAlVe gEnetic Research - BRAVE Study
Brief Title: The BRAVE Study- The Identification of Genetic Variants Associated With Bicuspid Aortic Valve Using a Combination of Case-control and Family-based Approaches.
Acronym: BRAVE
Status: Recruiting | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 165756
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and plasma to be retained at minus 80 degrees
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational

SUMMARY:
Bicuspid aortic valve (BAV) is the most common congenital heart anomaly in the general population (1-2% of all individuals). In affected people, the aortic valve (the structure ensuring one way blood flow between the heart's left pumping chamber, the left ventricle and the main body artery, the aorta) consists of 2 rather than 3 leaflets. This arrangement can cause the affected valve to have restricted opening or cause it to leak. Both situations put strain on the heart and patients with BAV across the age range may require surgery to replace the affected valve. BAV is therefore a condition associated with significant ill health and early mortality.

BAV is known to cluster in families and is likely to have a genetic cause. We don't fully understand the inheritance of BAV or the specific genes involved in its development. Learning more about this is the basis of the BRAVE study.

We will ask patients with BAV and their relatives (who may or may not have BAV) to take part in the study. Blood samples obtained from the participants will be used for analyses of their genetic composition. This information, linked with the clinical data concerning who does and does not have BAV, will potentially enable the identification of the gene changes responsible for the disease. This, we hope, will give us a much better understanding of the mechanisms leading to this serious and common condition.

DETAILED DESCRIPTION:
Bicuspid aortic valve is the most common congenital valvular heart anomaly in the general population, with a prevalence estimated between 0.5 - 2%. It is more common in males than females with ratios reported between 2:1 and 3:1. The prevalence of BAV shows significant differences amongst different ethnic groups. BAV sometimes associates with other, non-valvular cardiovascular phenotypes, e.g. aortic coarctation, left dominant coronary artery system and intracranial aneurysms. Presence of BAV is strongly associated with dilatation of the ascending aorta irrespective of valve function. BAV related dilatation of the ascending aorta has been reported in 56% of those aged 30 years old and 88% of those aged 80 years old.

Presence of BAV can be associated with serious cardiovascular complications. In a long term observational study, the overall survival of BAV patients was equal to age and sex matched subjects from the general population, but BAV was associated with the need for surgical intervention in 27% of subjects. Additionally, cardiovascular medical events (heart failure, infective endocarditis and stroke) occurred in 33% of all subjects with BAV over that period.

BAV shows strong familial clustering, indicating that it has a strong genetic basis. In an echocardiographic survey of first degree relatives of patients with BAV 36.7% of families had at least 2 members with this anomaly. In a study of 309 subjects from 48 extended families heritability of BAV was calculated at 89%.A whole genome linkage scan performed in 38 extended families (324 individuals), showed evidence for linkage with 5 chromosomal loci - 18q22, 5q21, 13q34, 9q34, 17q24. When analysed separately, the majority of families contributed only to a single locus suggesting heterogenic genetic origin of BAV. Based on these observation an oligogenic model of autosomal dominant inheritance with reduced penetrance has been suggested.

Despite strong familial clustering, only few genetic loci have been associated with BAV so far. The strongest evidence exist for association of BAV with NOTCH1 gene (translocation associated protein) - the product of which is an important element in developmental control of cell fate decisions. Other candidate loci include TGFBR2 (transforming growth factor beta receptor 2 gene), GATA5 (GATA-binding protein gene) and eNOS (endothelial nitric oxide synthase gene). However, the identified loci explain only small proportion of BAV heritability.

Modern DNA analysis, notably next generation sequencing, allows variants associated with disease to be identified more rapidly and with increased precision. The objective of this project is to use such technology to identify genetic variants and genes predisposing to BAV using a combination of case-control and family-based approaches. A better understanding of the genetic underpinnings of BAV could in the future help to improve the management of this valvular heart condition.

This BRAVE study will recruit patients with antecedent or new diagnosis of BAV. As many relatives of the index patient as possible will be recruited to the study (family based analysis). They will be screened with echocardiography for the presence of BAV. Additional group of unrelated healthy individuals with three leaflet valves will be recruited for the purpose of case control analysis.

Demographic and clinical data from all participants will be collected using purposefully designed questionnaires and by accessing their medical records. Data on imaging investigations will be obtained from the medical records or from the echocardiogram performed for the purpose of screening.

Blood samples will be used for the purpose of isolation of genetic material and subsequent genetic analysis. Additional laboratory tests may be performed on the blood samples to provide supporting evidence to the results of genetic analysis.

The main analyses will consist of identifying and cataloguing genetic variants for each individual from the DNA sequencing and then seeing whether any particular variant or sets of variants are more commonly present in BAV subjects versus those without BAV (case-control design) or present in subjects with BAV but not in unaffected family members (family-based approach).

ELIGIBILITY:
Inclusion Criteria:

- 1. All outpatients and inpatients with diagnosed BAV, of either gender, aged 10 and above.

2. Affected and unaffected first degree relatives meeting the age criteria.

Exclusion Criteria:

* 1) Patients unable to give informed consent.

  2) Patients known to be infected with HIV, Hepatitis B, Hepatitis C or any other agent posing an infection risk from unfixed material.

  3) Patient with known cytogenetic disorders e.g. aneuploidia, chromosomal abnormalities and known karyotype abnormalities.

  4) Patients with diagnosed or suspected Mendelian syndromes (e.g. Marfan syndrome, Loeys-Dietz syndrome, Ehlers-Danlos syndrome).

Ages: 10 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Suitable patients with the condition (index patients) will be identified and invited to take part in the study by their healthcare teams. Relatives will be identified during the interview with the index patient and invited to take part in the study by the index patients.
  Subjects below the age of 18 will be provided with age specific documents (information leaflets, invitation letters and consent forms). Informed consent will be sought from such participants as well as parent or legal guardian of such participants.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-09-08 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the BRAVE study is to identify genetic loci associated with BAV. | 48 Months
  The main analyses will consist of identifying and cataloguing genetic variants for each individual from the DNA sequencing and then seeing whether any particular variant or sets of variants are more commonly present in BAV subjects versus those without BAV (case-control design) or present in subjects with BAV but not in unaffected family members (family-based approach).

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Bolger, Dr, Principal Investigator — Principal Investigator
Locations (4):
- United Kingdom (4):
  - Kettering General Hospital, Kettering
  - University Hospitals of Leicester, Leicester
  - Imperial College Healthcare NHS Trust, London
  - Sheffield Teaching Hospital NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No